CLINICAL TRIAL: NCT03918538
Title: A Series of Study in Testing Efficacy of Pulmonary Rehabilitation Interventions in Lung Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 13MMHIS305
Record Dates: First submitted 2019-04-16; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
Keywords: lung cancer; early physical rehabilitation; muscle endurance; aerobic capacity; quality of life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): After pre-test, the intervention participants received a 60 minutes of teaching regarding the home rehabilitation exercise program, with a printed exercise manual.
  The intervention participants also received a weekly phone call from the interventionist to enhance their exercise adherence and helping to overcome exercise barriers.
  Interventions: Behavioral: Home rehabilitation exercise program
- The control group (No Intervention): Participants in the control group received regular medication education.

INTERVENTIONS:
Behavioral: Home rehabilitation exercise program — After pre-test, the intervention participants received a 60 minutes of teaching regarding the home rehabilitation exercise program, with a printed exercise manual. The intervention participants also received a weekly phone call from the interventionist to enhance their exercise adherence and helping to overcome exercise barriers.
  Arms: The intervention group

SUMMARY:
Aim: To develop and testing a home exercise program for lung cancer survivors to improve their exercise tolerance and quality of life during the rehabilitation phase.

Design: An experimental design will be used in the study. The 90 lung cancer survivors, who were diagnosed with lung cancer within one year and have completed their initial cancer treatment, will be recruited and randomized to the control or intervention group. After pre-test, the intervention participants will receive a 60 minutes of teaching regarding the home rehabilitation exercise program, with a printed exercise manual. The intervention participant will also receive a weekly phone call from the interventionist to enhance their exercise adherence and helping to overcome exercise barriers. The similar outcome measures as study one will be assessed on the baseline, 1th month, 3th month, and 6th month.

Measurements: The study outcomes will be evaluated by three physical measures, six-minute walk test, Modified Borg Scale, 30-second Chair Sit-to-Stand Test, and 30-second Chair Sit-to-Stand Test, as well as a study questionnaire including Functional Assessment of Cancer Therapy-Lung (FACT-L) and FACIT-Fatigue. For study one the following data will be collected from the patient'schart: post-operative pulmonary complications, days of chest tube insertion, and days of hospitalization.

Data analysis: Descriptive analysis will be used to describe patients'demongraphics, disease variables, and outcome variables. The Chi-square, T-test, and General Linear Mix-effect Model will be used to test the efficacy of the study interventions.

DETAILED DESCRIPTION:
Background: With appropriate treatment, lung cancer patients can be a long-term survivor. However, many patients suffered from post-operative pulmonary complications, limited activity tolerance, and poor quality of life. Nurses in a great position to provide individualized health education regarding exercise for these patients; therefore to develop and test cost-effective nurses-lead lung rehabilitation exercise education programs deserver further scientific efforts.

Aim: To develop and testing a home exercise program for lung cancer survivors to improve their exercise tolerance and quality of life during the rehabilitation phase.

Design: An experimental design will be used in the study. The 90 lung cancer survivors, who were diagnosed with lung cancer within one year and have completed their initial cancer treatment, will be recruited and randomized to the control or intervention group. After pre-test, the intervention participants will receive a 60 minutes of teaching regarding the home rehabilitation exercise program, with a printed exercise manual. The intervention participant will also receive a weekly phone call from the interventionist to enhance their exercise adherence and helping to overcome exercise barriers. The similar outcome measures as study one will be assessed on the baseline, 1th month, 3th month, and 6th month.

Measurements: The study outcomes will be evaluated by three physical measures, six-minute walk test, Modified Borg Scale, 30-second Chair Sit-to-Stand Test, and 30-second Chair Sit-to-Stand Test, as well as a study questionnaire including Functional Assessment of Cancer Therapy-Lung (FACT-L) and FACIT-Fatigue. For study one the following data will be collected from the patient'schart: post-operative pulmonary complications, days of chest tube insertion, and days of hospitalization.

Data analysis: Descriptive analysis will be used to describe patients'demongraphics, disease variables, and outcome variables. The Chi-square, T-test, and General Linear Mix-effect Model will be used to test the efficacy of the study interventions.

Significance: The study results will provide evidence for the efficacy of pulmonary rehabilitation and a home exercise program for enhancing exercise tolerance and quality of life in lung cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. aged 20 and older,
2. diagnosed with stage I-IIIB non-small cell lung cancer
3. completed initial cancer treatments and no planned cancer treatment in three months
4. Karnofsdy Performance Status equal or greater then 50
5. estimated survival time greater than six months
6. with the permission of the patient's physician

Exclusion Criteria:

1. having a medical condition precluding exercise (i.e. uncontrolled arrhythmias, uncontrolled hypertension, third-degree heart block, myocardial infarction within six months, unstable angina, acute congestive heart failure and taking anticoagulation for valve diseases).
2. poor controlled diabetics (HbA1C>9%)
3. regularly exercising in moderate or higher intensity three time a week within three month
4. unable to walk independently
5. unable to communicate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
six-minute walk test | Change from Baseline to 6 months
  The six-minute walk test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.

SECONDARY OUTCOMES:
30-second arm curl test | Change from Baseline to 6 months
  To measure upper body strength and endurance. The participant is sitting on the edge of a stabile chair, with seat height of 44 cm (originally 43.18 cm). The back is outstretched, the feet resting flat on the ground. A handle weighing 2 kg for women or 3.5 kg for men is held in the dominant hand. The arm is directed downwards, along the chair, perpendicularly to the floor. Participant's task is, at a command given by the testing person, to rotate the hand upwards while simultaneously flexing the extremity in the elbow (flexion with supination), and subsequently to extend the extremity to its baseline position.
30-second chair sit-to-stand test | Change from Baseline to 6 months
  To test leg strength and endurance. Record the number of stand a person can complete in 30 seconds.
Functional Assessment of Cancer Therapy-Lung (FACT-L) | Change from Baseline to 6 months
  There are two subscales, 27 items of FACT-General and 9 items of Lung Cancer Subscale. Each item is rated on a 5-point Likert scale (0-4). The total score of the 36 items represents the score of the scale. The higher values represent better quality of life.
The Functional Assessment of Chronic Illness Therapy-Fatigue | Change from Baseline to 6 months
  There are 13 items in the scale. Each item is rated on a 5-point Likert scale (0-4). The total score of the 13 items represents the score of the scale. The possible score for the scale ranges from 0 to 52. The higher values represent more fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Tsae Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benzo R, Wigle D, Novotny P, Wetzstein M, Nichols F, Shen RK, Cassivi S, Deschamps C. Preoperative pulmonary rehabilitation before lung cancer resection: results from two randomized studies. Lung Cancer. 2011 Dec;74(3):441-5. doi: 10.1016/j.lungcan.2011.05.011. Epub 2011 Jun 12. PMID 21663994
- [Background] Jones LW, Peddle CJ, Eves ND, Haykowsky MJ, Courneya KS, Mackey JR, Joy AA, Kumar V, Winton TW, Reiman T. Effects of presurgical exercise training on cardiorespiratory fitness among patients undergoing thoracic surgery for malignant lung lesions. Cancer. 2007 Aug 1;110(3):590-8. doi: 10.1002/cncr.22830. PMID 17582629
- [Background] Peddle CJ, Jones LW, Eves ND, Reiman T, Sellar CM, Winton T, Courneya KS. Effects of presurgical exercise training on quality of life in patients undergoing lung resection for suspected malignancy: a pilot study. Cancer Nurs. 2009 Mar-Apr;32(2):158-65. doi: 10.1097/NCC.0b013e3181982ca1. PMID 19258829